CLINICAL TRIAL: NCT02113579
Title: Assessment of a Potassium Oxalate Containing Formulation for the Relief of Dentinal Hypersensitivity
Brief Title: Test on a New Experimental Mouth Rinse for Relieving Tooth Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOXDHY0009
Record Dates: First submitted 2014-04-08; First posted 2014-04-14 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Dentin Sensitivity
Keywords: Tooth Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KOX (Experimental): After brushing for at least one-minute using at least one-inch strip of toothpaste, rinse with water and then rinse 60 seconds with 10mL of mouth rinse, twice daily.
  Fluoride Toothpaste / Crest® Cavity Protection Regular and Experimental Mouth Rinse 12027-033
  Interventions: Device: Experimental Mouth Rinse 12027-033
- PLA (Placebo Comparator): After brushing for at least one-minute using at least one-inch strip of toothpaste, rinse with water and then rinse 60 seconds with 10mL of mouth rinse, twice daily.
  Fluoride Toothpaste/Crest® Cavity Protection Regular and Placebo Mouth Rinse
  Interventions: Other: Placebo Mouth Rinse

INTERVENTIONS:
Device: Experimental Mouth Rinse 12027-033 — After brushing for at least one-minute using at least one-inch strip of toothpaste, rinse with water and then rinse 60 seconds with 10mL of mouth rinse, twice daily.
  Other Names: Fluoride Toothpaste / Crest® Cavity Protection Regular
  Arms: KOX
Other: Placebo Mouth Rinse — After brushing for at least one-minute using at least one-inch strip of toothpaste, rinse with water and then rinse 60 seconds with 10mL of mouth rinse, twice daily.
  Other Names: Fluoride Toothpaste/Crest® Cavity Protection Regular
  Arms: PLA

SUMMARY:
This study is for people with sensitive teeth and involves going to the dentist for 4 visits over 6 weeks. At each visit the dentist will look at the mouth, teeth, tongue and gums of participants, and check for sensitive teeth.

During the first 2 weeks, participants will brush their teeth 2 times a day with the fluoride toothpaste provided.

Then, if they qualify to continue in the study, participants will be assigned to one of two treatment groups for the last 4 weeks. Both groups will use assigned toothpaste currently sold on the market. Both groups will each have an investigative mouth rinse to use as well. Participants will have an equal chance of being assigned to any one of the three groups.

For the next 4 weeks, participants will use their assigned products according to the directions provided. At Visit 1, participants will be supervised while they brush their teeth to ensure they understand the directions. They will also have supervised use of the products at Visit 2.

Results will be analyzed to assess whether the mouthwashes help to reduce tooth sensitivity during the study.

DETAILED DESCRIPTION:
This study will consist of run-in and treatment phases. To qualify for the study, participants must meet the inclusion/exclusion criteria and return tactile sensitivity scores within protocol-specified parameters at both the screening and baseline visits.

Run-in will consist of a 2-week period during which participants will use a sodium fluoride dentifrice. At the start of the first phase, participants will attend a Screening Visit. They will participate in the informed consent process, complete a medical/dental history, and be evaluated for tactile sensitivity to Yeaple probe and response to a cold air stimulus.

Participants who qualify through screening will begin a run-in period that will last approximately two weeks. The run-in period will be followed by a Baseline visit. Participants who continue to qualify through Baseline will be randomly assigned to one of two treatment groups.

During the four-week treatment period, all participants will brush their teeth twice daily for at least one minute in their usual manner, with their assigned toothpaste. After brushing, participants will rinse with water, and then rinse with 10 mL of their assigned experimental mouth rinse for 60 seconds.

The study duration is approximately six weeks with each participant visiting the clinical site four times.

Adverse events will be observed and collected by querying each participant at each visit for new or continuing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age in good general and oral health without any known allergy to commercial dental products or cosmetics.
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the study
* Females of childbearing potential must be using a medically-acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the study. Acceptable methods for this study include:
* Abstinence
* Birth control pills, patches, vaginal rings, implants or injections
* Intrauterine device
* Double barrier method (condom/diaphragm or cervical cap with spermicide)
* Bilateral tubal ligation
* Hysterectomy
* Ovariectomy
* Male partner vasectomy
* Willingness to use the assigned products according to instructions, availability for appointments, and likelihood of completing the clinical study.
* A minimum of 2 natural premolars, canines, and/or incisors teeth with decay-free scorable facial/buccal surfaces which must present cervical abrasion, and/or erosion and/or gingival recession.
* A minimum of two eligible teeth (premolars, canines and/or incisors) with a Screening (-2 weeks Baseline) and Baseline cold air stimulus Visual Analogue Scale (VAS) score of 40 - 80 mm on a 100 mm VAS scale, tactile sensitivity score between 10 - 30 grams after application of the Yeaple probe and a tactile (Yeaple probe) VAS of 40 -80 mm on a 100 mm VAS scale.
* No more than two eligible teeth per quadrant each separated by 2 other teeth must be selected.
* Absence of significant oral soft tissue pathology, based on the dentist's visual examination and at the discretion of the investigator.
* Adequate oral hygiene (i.e. brush teeth daily and exhibit no signs of oral neglect).
* Absence of severe marginal gingivitis, moderate/advanced periodontitis (ADA Type III, IV) based on a clinical examination and discretion of the Investigator.
* Absence of extensive absence of extensive calculus above the gum line.

Exclusion Criteria:

* Volunteers who report history or presence of kidney disorders, kidney stones, have celiac disease, inflammatory bowel disease (ulcerative colitis or Crohn's disease), chronic pancreatitis, have had intestinal or weight-loss surgery, or if have stomach or intestinal problems that keep them from absorbing certain foods or nutrients.
* Volunteers with eating disorders, uncontrolled Gastroesophageal reflux disease GERD or Acid Reflux, excessive dietary or environmental exposure to acids, or other systemic conditions that are predisposing to dentinal hypersensitivity.
* Volunteers with chronic medical debilitating disease associated with constant or intermittent episodes of daily pain.
* Long-term daily use (≥ 7 consecutive days) of analgesics and any other drugs that at the discretion of the Investigator would compromise the response of the hypersensitivity assessments.
* Volunteers who have been using any home-care bleaching, whitening products or have had a professional bleaching treatment within 4 weeks of the Screening visit.
* Use of desensitizing agents whether prescribed or over-the-counter within eight weeks prior to screening visit (any sensitivity toothpastes such as Crest Sensitivity, Sensodyne, Crest Pro-Health, Colgate Sensitivity Relief, any mouthwash and oral care products used for the treatment of dentinal hypersensitivity).
* Volunteers who during the study will receive dental treatment which may affect their dentinal hypersensitivity condition (i.e., oral prophylaxis). Emergency treatment will be allowed.
* Those with a known allergy to study products' ingredients.
* Those requiring antibiotic premedication prior to invasive dental procedures.
* Participation in a dental clinical study involving oral care products within the past 30 days.
* Self reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results)
* Teeth that are grossly carious, orthodontically banded, abutment teeth for fixed or removable prostheses, crowned teeth, or third molars will not be included in the study.
* Periodontal surgery and orthodontic treatment within previous 3 months.
* Extensive restorative treatment (i.e. extensively restored teeth or teeth with restoration(s) extending into the test area) at the discretion of the Investigator.
* Dental prophylaxis within 2 weeks prior to Screening visit.
* Teeth or periodontium with pathology or defect likely to cause pain.
* Teeth with clinical mobility > grade 1.
* Relative, partner or staff of any clinical research site personnel
* Participation in any clinical study within 30 days of Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lynch, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (2):
- United States (2):
  - Salus Research, Inc., Fort Wayne, Indiana
  - Silverstone, Las Vegas, Nevada

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Control: Placebo Mouth Rinse (10 mL) twice daily after brushing
- 12027-033: Experimental Mouth Rinse 12027-033 (10 mL) twice daily after brushing
Period: Overall Study
Arm/Group | Placebo Control | 12027-033
Started | 186 | 189
Completed | 176 | 185
Not Completed | 10 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Control | 12027-033 | Total
Number analyzed (Participants) | 186 | 189 | 375
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (12.05) | 38.0 (12.03) | 38.5 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 145 | 283
  Male | 48 | 44 | 92
Region of Enrollment [Number; unit: participants]
  USA | 186 | 189 | 375

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Reduction From Baseline by at Least 30% in Mean Cold Air VAS Stimulus Score at Week 4
Description: Tooth sensitivity was measured using a Cold Air Stimulus. When being assessed, participants rated their perception of the pain/discomfort experienced when cold air was directed at the exposed root of each tooth by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The score for each participant was calculated by averaging the scores for all study teeth for that participant. A participant was considered an individual success if the participant's mean cold air stimulus VAS score at Week 4 was at least 30% lower than the participant's mean baseline cold air stimulus VAS score.
Time Frame: 4 Weeks
Population: Analysis was based on Full Analysis Set, which included all randomized subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
percentage of participants | 44.6 | 69.3
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; The null hypothesis was no difference in success rates between treatment groups. The alternative hypothesis was a difference in success rates between treatment groups; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Per statistical analysis plan, if experimental rinse was significantly better than placebo (p<0.05) with estimated difference of >= 20%, testing proceeded to Mean Cold Air Stimulus VAS Score at Week 4. Family-wise error was controlled at 0.05; Study center and mean baseline cold air stimulus VAS score as covariate. For subjects with no score at Week 4, non-response was imputed; Success rate difference (%) = 24.70 — Estimated by calculating the model predicted success probabilities assuming all subjects received 12027-033 and then assuming all subjects received placebo, and then calculating mean of subjects' differences between these predicted probabilities

2. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 4
Description: Tooth sensitivity was measured using a Cold Air Stimulus. When being assessed, participants rated their perception of the pain/discomfort experienced when cold air was directed at the exposed root of each tooth by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 4 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
units on a scale (mm) | 40.04 (1.597) | 25.76 (1.569)
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; The null hypothesis was no difference in mean outcome between treatment groups. The alternative hypothesis was a difference in mean outcome between treatment groups; Test type: Superiority or Other; p < 0.001, Repeated Measures Model — Per statistical analysis plan, if experimental rinse was significantly better than placebo (p<0.05), testing proceeded to Mean Tactile Sensitivity Score at Week 4. Family-wise error was controlled at 0.05; Analysis included Weeks 2 and 4 data. Terms included treatment, visit, study center, baseline value, treatment-by-visit and baseline-by-visit; Least Squares Mean Difference = -14.27, 95% CI 2-sided [-18.68 to -9.87], Standard Error of Mean 2.239 — For subjects without post-baseline data, the baseline value was carried forward to Week 2. An unstructured covariance pattern was assumed

3. Secondary Outcome: Mean Tactile Sensitivity Score at Week 4
Description: Tooth sensitivity was measured using a Yeaple probe. The force at which discomfort was felt by the participant was recorded on a scale of 10-80 grams. The score for each participant was calculated by averaging the scores for all study teeth for that participant, at each visit.
Time Frame: 4 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
grams | 15.29 (1.315) | 28.74 (1.292)
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures Model — Per statistical analysis plan, if experimental rinse was significantly better than placebo (p<0.05), testing proceeded to Mean Cold Air Stimulus VAS Score at Week 2 and Mean Tactile Sensitivity Score at Week 2. Family-wise error controlled at 0.05; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = 13.45, 95% CI 2-sided [9.83 to 17.08], Standard Error of Mean 1.844 — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Mean Cold Air Stimulus VAS Score at Week 2
Description: as for outcome 2
Time Frame: 2 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
units on a scale (mm) | 48.04 (1.284) | 40.37 (1.274)
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures Model — Per statistical analysis plan, Hochberg's method at significance level 0.05 was applied to jointly evaluate secondary outcomes Mean Cold Air Stimulus VAS Score at Wk 2 and Mean Tactile Sensitivity Score at Wk 2. Family-wise error controlled at 0.05; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.67, 95% CI 2-sided [-11.23 to -4.11], Standard Error of Mean 1.809 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Mean Tactile Sensitivity Score at Week 2
Description: as for outcome 3
Time Frame: 2 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
grams | 12.72 (0.692) | 17.42 (0.687)
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures Model — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = 4.70, 95% CI 2-sided [2.78 to 6.62], Standard Error of Mean 0.975 — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Percentage of Subjects With Reduction From Baseline by at Least 30% in Mean Cold Air VAS Stimulus Score at Week 2
Description: Tooth sensitivity was measured using a Cold Air Stimulus. When being assessed, participants rated their perception of the pain/discomfort experienced when cold air was directed at the exposed root of each tooth by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The score for each participant was calculated by averaging the scores for all study teeth for that participant. A participant was considered an individual success if the participant's mean cold air stimulus VAS score at Week 2 was at least 30% lower than the participant's mean baseline cold air stimulus VAS score.
Time Frame: 2 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
percentage of participants | 30.6 | 46.0
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; Study center and mean baseline cold air stimulus VAS score as covariate. For subjects with no score at Week 2, non-response was imputed; Success rate difference (%) = 15.44 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 2
Description: Tooth sensitivity was measured using a Visual Analogue Scale (VAS). At each visit, participants rated their perception of the pain/discomfort experienced from the Yeaple probe by marking a single vertical line on a VAS scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm. The investigator recorded a VAS score of 0 mm for participants who did not experience discomfort at the maximum force of 80 grams. The score for each participant was calculated by averaging the scores for all study teeth for that participant.
Time Frame: 2 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
units on a scale (mm) | 44.39 (1.170) | 37.72 (1.161)
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures Model — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.67, 95% CI 2-sided [-9.92 to -3.43], Standard Error of Mean 1.650 — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Mean Tactile Sensitivity VAS Score at Week 4
Description: as for outcome 7
Time Frame: 4 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
units on a scale (mm) | 38.24 (1.368) | 26.72 (1.345)
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures Model — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -11.52, 95% CI 2-sided [-15.30 to -7.75], Standard Error of Mean 1.920 — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Global Subjective VAS Score at Week 2
Description: At each visit, participants rated their perception of the pain/discomfort experienced by marking a single vertical line on a Visual Analogue Scale (VAS) scale from 0 to 100 mm, where 0 = No Pain/Discomfort and 100 = Intense Pain/Discomfort. Participants were instructed as follows:"Please rate the intensity of the pain/discomfort you have experienced in the last two weeks when drinking cold/hot beverages and/or foods, eating sweet and sour foods, breathing cold air, brushing your teeth or performing any habits/behaviors that elicit your dentinal hypersensitivity pain/discomfort since you have been using the product." The dental recorder measured the length of the line from 0 to the participant's line and recorded the VAS score in mm.
Time Frame: 2 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
units on a scale (mm) | 45.33 (1.009) | 42.09 (1.001)
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.023, Repeated Measures Model — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.24, 95% CI 2-sided [-6.04 to -0.45], Standard Error of Mean 1.422 — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Global Subjective VAS Score at Week 4
Description: as for outcome 9
Time Frame: 4 Weeks
Population: Analysis was based on the Full Analysis Set, which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale (mm)
Arm/Group | Placebo Control | 12027-033
Number analyzed (Participants) | 186 | 189
units on a scale (mm) | 39.00 (1.337) | 31.39 (1.311)
Statistical Analysis 1: Comparison: Placebo Control vs 12027-033; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Repeated Measures Model — The significance threshold level was 0.05 (two-sided), with no multiple comparisons adjustment; [statistical method as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.61, 95% CI 2-sided [-11.29 to -3.93], Standard Error of Mean 1.873 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Day 28 ± 3 days, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 4 (Day 28 ± 3 days). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Placebo Control | 12027-033
Serious Adverse Events (participants affected / at risk) | 0/186 | 0/189
Other Adverse Events (participants affected / at risk) | 0/186 | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators agreed not to publish the study results without prior sponsor approval.